CLINICAL TRIAL: NCT06073574
Title: The CARDIO-TTRansform Magnetic Resonance Imaging (MRI) Sub-study
Brief Title: CARDIO-TTRansform Magnetic Resonance Imaging (MRI) Sub-study
Status: Active, not recruiting | Type: Observational
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ION-682884-CS2MRI; 2019-002835-27 (EudraCT Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR-CM)
Keywords: TTR; Amyloidosis; Cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Experimental: ION-682884-CS2 MRI Scan Sub-set: Participants enrolled in the parent study ION-682884-CS2 (NCT04136171) to receive either eplontersen or placebo and who consented to participate in this sub-study will undergo cardiac MRI at Baseline, Weeks 25, 49, 97 and 140.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — MRI Scans as specified in the corresponding arm group.

SUMMARY:
The main purpose of this study is to measure the amyloid burden, defined as extracellular volume (ECV) assessed by Magnetic Resonance Imaging (MRI) over time in a subset of up to 150 participants enrolled in ION-682884-CS2 (NCT04136171).

DETAILED DESCRIPTION:
This pilot study will determine the efficacy of ION-682284 in reducing the amyloid deposit on the heart tissue compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

To participate in the ION-682884-CS2MRI sub-study, participants must meet all inclusion criteria of the study protocol ION-682884-CS2 (NCT04136171).

Exclusion Criteria

1. Contraindication or sensitivity to MRI contrast agents
2. Orthopnea of sufficient severity to preclude supine scanning at screening.
3. Weight or body girth exceeds the limits of the cardiac MRI machine specifications.
4. Contraindication to cardiac MRI scanning, as assessed by local MRI safety questionnaire/checklist.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were randomized in Study ION-682884-CS2 (NCT04136171) and who signed informed consent for the MRI sub-study will participate in this sub-study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in the Percent of ECV in Participants Receiving ION-682884 vs. Placebo According to ION-682884-CS2 Treatment Groups | From Baseline up to Week 140

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Oregon Health and Science University, Portland, Oregon
- Italy (2):
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Azienda Ospedale Università di Padova, Padua
- Hospital Universitario Puerta de Hierro, Majadahonda, Spain
- United Kingdom (6):
  - Synexus - Scotland Clinical Research Centre, Bellshill
  - Synexus Midlands Clinical Research Centre, Birmingham
  - Synexus - Wales, Cardiff
  - Royal Free London NHS Foundation Trust, London
  - Richmond Pharmacology, London
  - Synexus - Manchester Clinical Research Centre, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CARDIO-TTransform Website — https://www.cardio-ttransform.com/